CLINICAL TRIAL: NCT05986578
Title: Identifying Electrophysiological Targets for Transcranial Magnetic Stimulation in Cocaine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Heather E. Webber, PhD, Instructor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSC-MS-21-0813 (Main study); K01DA058765 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cocaine Use Disorder
Keywords: Transcranial Magnetic Stimulation (TMS); Event-Related Potentials; Substance Use Disorder; Reward Positivity; Late Positive Potential
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- dlPFC then dmPFC then Sham iTBS (Experimental)
  Interventions: Device: TMS to dmPFC; Device: TMS to dlPFC; Device: Sham iTBS
- dmPFC then dlPFC then sham iTBS (Experimental)
  Interventions: Device: TMS to dmPFC; Device: TMS to dlPFC; Device: Sham iTBS
- dmPFC then sham iTBS then dlPFC (Experimental)
  Interventions: Device: TMS to dmPFC; Device: TMS to dlPFC; Device: Sham iTBS
- dlPFC then sham iTBS then dmPFC (Experimental)
  Interventions: Device: TMS to dmPFC; Device: TMS to dlPFC; Device: Sham iTBS
- sham iTBS then dlPFC then dmPFC (Experimental)
  Interventions: Device: TMS to dmPFC; Device: TMS to dlPFC; Device: Sham iTBS
- shami iTBS then dmPFC then dl PFC (Experimental)
  Interventions: Device: TMS to dmPFC; Device: TMS to dlPFC; Device: Sham iTBS

INTERVENTIONS:
Device: TMS to dmPFC — TMS will be delivered with a MagVenture Mag Pro R30 with the Cool-B70 A/P coil with active liquid cooling and active/sham sides. For dmPFC, approximately 25% of the nasion-inion distance or Talairah coordinates X 0 Y+60 Z+60 will be measured. The first session will begin with the acquisition of the resting motor threshold (rMT) on the contralateral hand. iTBS (triplet 50 Hz bursts, repeated at 5 Hz, 2 sec on and 8 sec off; 600 pulses per session) will be delivered at 110% of the rMT and will last ~3 minutes. The stimulation will start at a lower percentage and ramp up over time to acclimate participant to the feeling of stimulation. The intensity will be lowered in participant cannot tolerate the stimulation. Each participant will receive 3 sessions per visit with a 15-20 minute interval between sessions to increase the likelihood of detecting acute effects.
Device: TMS to dlPFC — TMS will be delivered with a MagVenture Mag Pro R30 with the Cool-B70 A/P coil with active liquid cooling and active/sham sides. For dlPFC, position F3 will be measured, using probabilistic EEG placement. The first session will begin with the acquisition of the resting motor threshold on the contralateral hand. iTBS (triplet 50 Hz bursts, repeated at 5 Hz, 2 sec on and 8 sec off; 600 pulses per session) will be delivered at 110% of the rMT and will last 3 minutes. The stimulation will start at a lower percentage and ramp up over time to acclimate participant to the feeling of stimulation. The intensity will be lowered in participant cannot tolerate the stimulation. Each participant will receive 3 sessions per visit with a 15-20 minute interval between sessions to increase the likelihood of detecting acute effects.
Device: Sham iTBS — Sham TMS will be delivered with the sham side of the MagVenture Cool B70 A/P coil. The software will be pre-programmed by a staff member that will not be involved in data analysis or collection for blinding purposes. The sham stimulation will match the number of pulses and length of time as the active condition and each participant will receive 3 sessions with a 15-20 min interval between sessions.

SUMMARY:
The purpose of this study is to assess effects of intermittent theta burst stimulation (iTBS) to left dorsolateral prefrontal cortex (dlPFC) and dorsomedial prefrontal cortex (dmPFC) compared to sham on electrophysiological indices of reward sensitivity and motivated attention in adults with cocaine use disorder.

ELIGIBILITY:
Inclusion Criteria:

* non-treatment-seeking adults
* meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for current cocaine use disorder of at least moderate severity (≥ 4 symptoms)
* have at least 1 positive urine Benzoylecgonine (BE) specimen (≥ 300 ng/mL) during intake
* be able to understand the consent form and provide written informed consent
* be able to provide the following verifiable information for a minimum of 2 contact persons: full legal name,email address, local mailing address, and as applicable, home, work, and cell phone numbers

Exclusion Criteria:

* current DSM-5 diagnosis for substance use disorder (of at least moderate severity) other than cocaine, marijuana, or nicotine
* in the opinion of the principal investigator (PI), the presence of any medical, neurological, psychiatric, or physical condition, disease, or illness that, may: (a) compromise interfere, limit, effect or reduce the subject's ability to complete the study; or (b) adversely impact the safety of the subject or the integrity of the data
* has current or recent (within 3 months of potential enrollment) suicidal ideation, suicidal behavior, homicidal ideation or a homicidal plan sufficient to raise subject safety concerns based on the following assessments according to the PI:

  1. Structured Clinical Interview for DSM-5 (SCID-5)
  2. Columbia Suicide Severity Rating Scale (C-SSRS) Screener - Answers YES to Questions 3, 4, 5, or 6
  3. Assault & Homicidal Danger Assessment Tool - Key to Danger > 1
* medical implants contraindicating TMS (i.e., aneurysm clips or coils, stents, implanted stimulators, implanted vagus nerve or deep brain stimulators, implanted electrical devices such as pacemakers or medication pumps electrodes for monitoring brain activity, cochlear implants for hearing, any magnetic implants, bullet fragments, any other metal device or object implanted in your body closer than 30 cm from the coil)
* history of brain surgery
* history of an intracranial lesion or any medical or neurological diagnosis/condition associated with increased intracranial pressure (i.e., Idiopathic Intracranial Hypertension/Pseudotumor Cerebri) OR any of the following symptoms within 30 days of enrollment: headaches > 15 days/month, loss of vision or decreased vision
* moderate-to-severe heart disease
* history of stroke
* is taking any antidepressant or antipsychotic medication at a dose above the maximum recommended dose or at a dose deemed to be potentially unsafe according to the PI; has taken any of the following medications, which are known to increase the risk of seizures, within 1 week of study enrollment; or does not agree to abstain from taking the following medications during study participation:

  1. clozapine137
  2. chlorpromazine137
  3. bupropion
  4. clomipramine hydrochloride
  5. amoxapine
  6. maprotiline hydrochloride
  7. diphenhydramine
  8. stimulants other than cocaine including the following:

     1. Dextroamphetamine and amphetamine
     2. Dextroamphetamine
     3. Lisdexamfetamine dimesylate
     4. Methamphetamine
     5. Methylphenidate
  9. tramadol
  10. isoniazid
* having conditions of probation or parole requiring reports of drug use to officers of the court
* personal history of epilepsy or seizure disorder and/or family history including a first-degree relative
* serious head injury with loss of consciousness
* impending incarceration
* pregnant or nursing for female patients
* inability to read, write, or speak English
* for adolescent aged participants (18-21 only): any risk factor for neurocardiogenic syncope (history of syncope/presyncope related to noxious stimuli, anxiety, micturition, or posture)
* hair style that is incompatible with EEG nets

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the amplitude of the Reward Positivity (RewP) component in microvolts in response to feedback on the Doors Task | Baseline(before iTBS session),immediately after iTBS session
  The Doors Task will be used to elicit the RewP component, representing reward sensitivity. The task is a guessing game, where participants guess which door contains a reward behind it. After selecting a door, the participants are notified if they found the prize by a green arrow pointing up or if they did not find the prize by a red arrow pointing down.
Change in the amplitude of the Late Positive Potential (LPP) in microvolts in response to visual stimuli on the Picture Viewing Task. | Baseline(before iTBS session),immediately after iTBS session
  The Picture Viewing Task will be used to elicit the LPP, reflecting the motivational salience of a stimulus. During this task, participants are asked to view a slide show of images including pleasant, unpleasant, neutral, and cocaine-related images.

SECONDARY OUTCOMES:
Change in craving as assessed by the Minnesota Cocaine Craving Scale (MCCS) | Baseline(before iTBS session),immediately after iTBS session
  The intensity of craving score will be used, scored from 1(none at all) to 10 (a great deal).
Change in pain as assessed by the Visual Analogue Scale | Baseline(before iTBS session),immediately after iTBS session
  This is scored from 1(no pain) to 10 (worst pain)
Change in cognitive function as assessed by the The Montreal Cognitive Assessment (MoCA) | Baseline(before iTBS session),immediately after iTBS session
  Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome.
Change in behavioral reward learning as assessed by the Pavlovian Go/No-Go task | Baseline(before iTBS session),immediately after iTBS session
  In the first "learning" phase, participants learn whether to press a button or withhold a response to receive a monetary reward or avoid a loss. In the second "transfer" phase, participants perform a forced choice task, where each of the predictive cues in the learning phase are paired with each other. Participants must select the "most rewarding" cue.
Change in Anhedonia as assessed by the Snaith Hamilton Pleasure Scale (SHAPS) | Baseline(before iTBS session),immediately after iTBS session
  This is a 14 item questionnaire. 9 of the questions are scored from 0(strongly disagree) to 3( strongly agree) and the rest are reverse coded with answer choices as follows: definitely agree, agree, disagree, and strongly disagree. Final scores range from 0-14 and higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Webber, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No